CLINICAL TRIAL: NCT03588715
Title: Pilot Study on Innate Activation and Viral Control in HIV-Infected Adults Undergoing an Analytical Treatment Interruption After Administration of Pegylated Interferon Alpha 2b With Broadly HIV-1 Neutralizing Antibodies (3BNC117, 10-1074)
Brief Title: Peg-Interferon Alpha 2b Combined With Two Intravenous Broadly HIV-1 Neutralizing Antibodies 3BNC117 and 10-1074 (BEAT-2)
Acronym: BEAT-2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Luis Montaner (Other)
Collaborators: University of Pennsylvania (Other); Philadelphia Fight (Other); Rockefeller University (Other); Merck Sharp & Dohme LLC (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Luis Montaner, Principal Investigator, The Wistar Institute
Organization: The Wistar Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES 38445; UM1AI126620 (NIH)
Record Dates: First submitted 2018-04-30; First posted 2018-07-17 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2020-06

CONDITIONS: HIV; HIV/AIDS; HIV-1 Infection
Keywords: HIV; HIV/AIDS; HIV Cure; HIV-1; HIV-1 Infection; BEAT-HIV; bNAbs; Broadly neutralizing antibodies
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — peginterferon alfa-2b; Broadly Neutralizing Antibodies

STUDY DESIGN:
Intervention Model Description: The study will evaluate the impact of the combination of 3BNC117 and 10-1074 with or without antiretroviral therapy in virological rebound during an ATI and effects on the HIV reservoir.
  This will be a pilot phase I study to evaluate the safety, tolerability, pharmacokinetics (PK), and antiviral activity of a combination of Pegylated Interferon alpha 2b with the two broadly neutralizing antibodies (3BNC117 and 10-1074) in 14 (all recruited first) individuals or the combination the broadly neutralizing antibodies alone in 7 (only 1 was able to be recruited due to COVID delays and drug availability) HIV-1 infected individuals, undergoing a brief analytical treatment interruption (ATI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegylated Interferon alpha 2b + bNAbs (Experimental): Pegylated Interferon alpha 2b (peg-IFN-α2b) + bNAbs (3BNC117 + 10-1074)
  Interventions: Drug: Pegylated Interferon alpha 2b (peg-IFN-α2b); Drug: 3BNC117 + 10-1074
- bNAb only (Experimental): bNAb (3BNC117 + 10-10-74) only
  Interventions: Drug: 3BNC117 + 10-1074

INTERVENTIONS:
Drug: Pegylated Interferon alpha 2b (peg-IFN-α2b) — Pegylated Interferon alpha 2b (peg-IFN-α2b) will be administered weekly via subcutaneous route.
  Other Names: Pegintron
  Arms: Pegylated Interferon alpha 2b + bNAbs
Drug: 3BNC117 + 10-1074 — Broadly Neutralizing Antibodies - Sequential, separate IV infusions of 3NBC117 + 10-1074.
  Other Names: Broadly Neutralizing Antibodies

SUMMARY:
This study will evaluate the safety, tolerability and innate immune mechanisms activation following administration of the combination of Pegylated Interferon alpha 2b (peg-IFN-α2b) with two broadly neutralizing antibodies (3BNC117 and 10-1074) in the setting of well-controlled HIV infection with antiretroviral treatment and a monitored analytical treatment interruption. The current proposal builds on previous experience using interferon alpha, 3BNC117 and 10-1074 alone in separate clinical trials that included a closely monitored analytical treatment interruption. The hypothesis is that the joint administration of peg-IFN-α2b with 3BNC117 and 10-1074 will be more effective than either intervention separately in suppressing HIV viremia during 8 weeks of analytical treatment interruption (Step 4) and reducing integrated HIV DNA in blood and tissue when measured during an analytical treatment interruption in patients with well-controlled HIV infection.

DETAILED DESCRIPTION:
The proposed study will evaluate the safety, tolerability and innate immune mechanisms activation following administration of the combination of Pegylated Interferon alpha 2b (peg-IFN-α2b) with two broadly neutralizing antibodies (3BNC117 and 10-1074) in the setting of well controlled HIV infection with antiretroviral treatment and a monitored analytical treatment interruption. This proposal builds on previous experience using interferon alpha, 3BNC117 and 10-1074 alone in separate clinical trials that included a closely monitored analytical treatment interruption. The hypothesis is that the joint administration of peg-IFN-α2b with 3BNC117 and 10-1074 will be more effective than either intervention separately in suppressing HIV viremia during 8 weeks of analytical treatment interruption (Step 4) and reducing integrated HIV DNA in blood and tissue when measured during an analytical treatment interruption in participants with well-controlled HIV infection. A review of the conceptual framework for the strategy to be tested includes:

* Why peg-IFN-α2? The therapeutic effects of peg-IFN-α2 yield two essential outcomes that are the fundamental objectives of HIV curative strategies: control viral replication in the absence of ART and reduce the levels of integrated HIV DNA in CD4+ T-cells. To date, peg-IFN-α is the only intervention that has been shown to maintain viral suppression to levels <50 copies/mL in the absence of ART in chronic infection. Preliminary data supports that correlates of anti-HIV reductions are centered on activation of NK responses.
* Why bNAbs + peg-IFN-α2b? The addition of bNAbs may act independently to control virus replication or decrease fitness thereby increasing the potential for a larger antiviral effect after IFN by enhance NK-mediated clearance via a reduced viral levels and the complementarity of bNAbs in enhancing mechanisms of antibody-mediated cytotoxicity against infected cells by binding to virus emerging from or viral proteins expressed on activated latent cells.
* Why combined bNAbs? In vivo, multiple bNAbs targeting different epitopes provide better neutralization and antigen recognition than single bNAbs, which suggests that adoptive transfer of multiple bNAbs may lead to superior viral control. Although bNAbs may have neutralization effects that are of greater clinical impact than ADCC, it is possible that antigen targeting through multiple bNAbs may also enhance NK-mediated cytotoxicity more than a single bNAb. The administration of broadly neutralizing antibodies alone in the setting of an analytical treatment interruption delays the return of viremia in a fraction of the participants.
* Why test an ATI of immunotherapy? To date, peg-IFN-α2 administered prior to an ATI or ART and subsequently maintained throughout the ATI period has maintained viral suppression. An effective curative strategy requires that all interventions be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA VL
* Ability and willingness of participant to provide informed consent
* Men and women aged ≥18 years
* Clinically stable on their first or second ART regimen that includes a boosted protease inhibitor or an integrase inhibitor. The current regimen should be stable for 4 weeks at the time of entry. Changes while the patient HIV viral load is undetectable does not count toward the number of ART regimens used, (for example an individual switching from an NNRTI-based regimen to an integrase inhibitor based regimen while the HIV viral load is undetectable will still be in their first regimen)
* HIV-1 RNA that is <50 copies/mL using a FDA-approved assay performed by any laboratory that has a CLIA certification or its equivalent within 56 days prior to study entry

NOTE: HIV-1 RNA must be measured at least once in the 24 weeks prior to entry and at least 3 days before the screening measure. Single determinations that are between ≥50 and <400 copies/mL (i.e., blips) are allowed as long as the preceding and subsequent determinations are <50 copies/mL. The screening value may serve as the subsequent determination <50 copies/mL following a blip

* Screening CD4+ T-cell count ≥450 cells/μL within 45 days prior to study entry
* Willingness to have blood samples collected and used for study-related research purposes
* The following laboratory values obtained within 45 days prior to enrollment:

  * Absolute neutrophil count (ANC) ≥1000 cells/mm3
  * Hemoglobin ≥12.0 g/dL for men and ≥11 g/dL for women
  * Platelet count 100,000/mm3
  * Creatinine clearance ≥60 mL/min estimated by the Cockcroft-Gault equation
  * Alanine aminotransferase (ALT) ≤2.5 x ULN
  * Pancreatic amylase ≤ 1.5 ULN and lipase ≤ 1.5 ULN and triglycerides ≤ 750 mg/dl
  * total bilirubin ≤ 1.5x ULN, (if not receiving atazanavir) OR direct bilirubin ≤ 1 mg/dl (if receiving atazanavir)
* For females of reproductive potential (i.e., women who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy), negative urine pregnancy test (with a sensitivity of 15-25 mIU/mL) within 48 hours prior to screening and entry.

ADDITIONAL REQUIREMENTS BIOLOGICAL FEMALES ARE NOTED IN CLINICAL PROTOCOL.

-Female partners of reproductive potential of male study participants on study drug would be educated that:

At least two of the following contraceptives MUST be used appropriately by female partners of reproductive potential of male study participants and/or their male partners with one method being highly effective and the other method being either highly effective or less effective as listed below:

Highly Effective Methods of Contraception

* Male condoms with spermicide
* Hormone-based contraceptives including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena by male participant's female partner of reproductive potential.
* Nonhormonal IUDs, such as ParaGard
* Tubal ligation
* Complete Abstinence*
* *Complete abstinence as defined as complete avoidance of heterosexual intercourse. Participants who choose complete abstinence are not required to use a second method of contraception. Acceptable alternate methods of highly effective contraception must be discussed in the event that the participant chooses to forego complete abstinence.

NOTE: Female partners of male participants participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug.

* Negative HBsAg result obtained within 6 months prior to study entry.
* HCV antibody negative result within 6 months prior to entry, or if the HCV antibody result is positive, a negative HCV RNA obtained within 6 months prior to study entry. Treated and cured HCV infected participants are allowed.
* Adequate venous access in at least one arm
* Body weight ≥ 125 and ≤ 300 lbs
* A non-clinically significant electrocardiogram (EKG, see section 7.2) for:

  1. men >45 years or women > 55 years of age
  2. younger subjects of either sex with two risk factors for coronary artery disease [smoking, hypertension (BP >140/90 or on antihypertensive medications), low HDL (<40 mg/dl), family history of premature CHD (<55 yrs males/<65 females
  3. subjects with a Framingham score > 15% (men) or 10% (women)

Exclusion Criteria:

* Susceptibility to bNAb 10-1074 based on IC90 greater than 2.0 µg/mL or susceptibility to bNAb 3BNC117 based on IC90 greater than 1.5 µg/mL using the Monogram Phenosense Assay on sample obtained on ART in absence of a subsequent documentation of a HIV viral load of greater than 1,000 copies on a collection date after that of the bNAb sensitivity sample.
* Previous receipt of humanized or human monoclonal antibody whether licensed or investigational
* Weight >300 lbs or <125 lbs
* History of an AIDS-defining illness
* Ongoing AIDS-related opportunistic infection (including oral thrush)
* History of a severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis in the 2 years prior to enrollment
* Currently pregnant, breastfeeding, or planning pregnancy
* Receipt of other investigational study agent within 30 days prior to enrollment
* Current or prior medications:

  * Confirmed clinical history of developing resistance to ART regimens that resulted in treatment changes
  * Receiving didanosine as part of the participant's ART regimen at the time of screening
  * Ongoing treatment with Isoniazid, Pyrazinamide, Rifabutin, Rifampicin, Ganciclovir, Valgancyclovir, Oxymetholone, Thalidomide or Theophylline.
  * Ongoing treatment with anticoagulants
  * Use of any investigational drug within 30 days prior to screening
  * History or current use of immunomodulatory therapy for over 2 weeks during the 6 months prior to enrollment, including, but not limited to:

    * IFN-α or γ (recombinant or pegylated)
    * Systemic corticosteroids (inhaled steroids allowed at the discretion of the Investigator)
    * Systemic cancer chemotherapy/irradiation
    * cyclosporin; tacrolimus (FK-506)
    * OKT-3
    * Any Interleukin, including IL-2
    * Cyclophosphamide
    * Methotrexate
    * IVIG (gamma globulin)
    * G/M-CSF
    * Hydroxyurea
    * Thalidomide
    * Pentoxifylline
    * Thymopentin, thymosin
    * Dithiocarbonate
    * Polyribonucleoside.
* History of adverse or allergic reactions to any type-1 interferon (e.g. IFN-α2a, IFN-α2b, IFN-β)
* Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer, including, clinically significant forms of:

  * Drug or alcohol abuse
  * Severe asthma
  * Uncontrolled hypertension
  * Type I diabetes mellitus, or type II diabetes mellitus that is not controlled with oral agents and/or insulin (i.e.: subjects with a history of diabetes mellitus and HA1C of > 9 in the last 3 months or at screening)
  * Psychiatric disorders, including severe depression and/or suicidal ideation
  * Heart disease
  * Cancer or hematologic malignancies
  * Prior diagnosis of multiple sclerosis or other neurodegenerative disorders
  * Liver cirrhosis or hepatic decompensation
  * Chronic HCV infection (HCV viremia), or HBV Ag positive and/ or HBV viremia (Notice: subjects with prior HCV infection with a documented sustained virologic response at 24 weeks post treatment prior to screening are eligible for enrollment.
  * Major organ transplantation with an existing functional graft
  * Active autoimmune diseases, including autoimmune hepatitis
  * History of retinopathy or clinically significant ophthalmologic disease
  * Opportunistic infections or other active infectious diseases
* Other conditions, such as active drug/alcohol abuse or dependence, that in the opinion of the Investigator would interfere with study compliance.
* Initiation of treatment during acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events during 30 week period of immunotherapy [Safety outcome] | 30 weeks of immunotherapy
  Number of participants with treatment-related adverse events during 30 weeks of peg-IFN-α2b administered at a weight adjusted dose weekly in combination with 3BNC117 and 10-1074 or the antibody combination alone.
Association between antibody-mediated cell cytotoxicity (ADCC) and NK cell activation as measured by flowcytometry at start of step 4 therapy interruption and level of HIV plasma viral load 8 week later [Innate Activation outcome] | 8 weeks after end of 30 week of immunotherapy (Analytical Treatment Interruption)
  Level of antibody-mediated cell cytotoxicity (ADCC) by direct measurement of NK cell CD107 degranulation against gp-120 coated targets in the presence of autologous plasma, and NK cell activation as measured by flowcytometry for frequency of cell subsets at start of step 4 therapy interruption. Values for ADCC cytotoxicity and NK activation will be tested by Spearman correlation test estimates with frequency of participants at <50 during the end of immune treatment Interruption (Step 4)
Frequency of subjects with plasma viral load <50 copies/ml after end of step 4 after ART therapy interruption [Virological outcome] | 8 weeks after end of 30 week of immunotherapy (Analytical Treatment Interruption)
  Frequency of participants remaining off ART with suppressed viral load (<50 copies/ml) at 8 weeks after immune therapy interruption.

CONTACTS AND LOCATIONS:
Overall Officials: Luis J Montaner, DVM, DPhil, Principal Investigator — The Wistar Institute; Pablo Tebas, M.D., Study Chair — University of Pennsylvania; Karam Mounzer, M.D., Study Director — Philadelphia Fight
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Jonathan Lax Center at Philadelphia FIGHT, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azzoni L, Foulkes AS, Papasavvas E, Mexas AM, Lynn KM, Mounzer K, Tebas P, Jacobson JM, Frank I, Busch MP, Deeks SG, Carrington M, O'Doherty U, Kostman J, Montaner LJ. Pegylated Interferon alfa-2a monotherapy results in suppression of HIV type 1 replication and decreased cell-associated HIV DNA integration. J Infect Dis. 2013 Jan 15;207(2):213-22. doi: 10.1093/infdis/jis663. Epub 2012 Oct 26. PMID 23105144
- [Background] Caskey M, Schoofs T, Gruell H, Settler A, Karagounis T, Kreider EF, Murrell B, Pfeifer N, Nogueira L, Oliveira TY, Learn GH, Cohen YZ, Lehmann C, Gillor D, Shimeliovich I, Unson-O'Brien C, Weiland D, Robles A, Kummerle T, Wyen C, Levin R, Witmer-Pack M, Eren K, Ignacio C, Kiss S, West AP Jr, Mouquet H, Zingman BS, Gulick RM, Keler T, Bjorkman PJ, Seaman MS, Hahn BH, Fatkenheuer G, Schlesinger SJ, Nussenzweig MC, Klein F. Antibody 10-1074 suppresses viremia in HIV-1-infected individuals. Nat Med. 2017 Feb;23(2):185-191. doi: 10.1038/nm.4268. Epub 2017 Jan 16. PMID 28092665
- [Background] Scheid JF, Horwitz JA, Bar-On Y, Kreider EF, Lu CL, Lorenzi JC, Feldmann A, Braunschweig M, Nogueira L, Oliveira T, Shimeliovich I, Patel R, Burke L, Cohen YZ, Hadrigan S, Settler A, Witmer-Pack M, West AP Jr, Juelg B, Keler T, Hawthorne T, Zingman B, Gulick RM, Pfeifer N, Learn GH, Seaman MS, Bjorkman PJ, Klein F, Schlesinger SJ, Walker BD, Hahn BH, Nussenzweig MC, Caskey M. HIV-1 antibody 3BNC117 suppresses viral rebound in humans during treatment interruption. Nature. 2016 Jul 28;535(7613):556-60. doi: 10.1038/nature18929. Epub 2016 Jun 22. PMID 27338952
- [Derived] Bilger A, Plenn E, Barg FK, Rendle KA, Carter WB, Lamour-Harrington A, Jones N, Peterson B, Sauceda JA, Tebas P, Mounzer K, Metzger D, Montaner LJ, Dube K. Participant experiences in HIV cure-directed trial with an extended analytical treatment interruption in Philadelphia, United States. HIV Res Clin Pract. 2023 Oct 6;24(1):2267825. Epub 2023 Oct 14. PMID 37837376
- [Derived] Neergaard R, Jones NL, Roebuck C, Rendle KA, Barbati Z, Peterson B, Tebas P, Mounzer K, Metzger D, Montaner LJ, Dube K, Barg FK. "I Know That I Was a Part of Making a Difference": Participant Motivations for Joining a Cure-Directed HIV Trial with an Analytical Treatment Interruption. AIDS Res Hum Retroviruses. 2023 Aug;39(8):414-421. doi: 10.1089/AID.2022.0040. Epub 2022 Sep 15. PMID 35979886
- See also: Website for the BEAT-HIV Delaney Collaboratory, which is the funding mechanism for the clinical trial outlined in the current registry. — http://beat-hiv.org